CLINICAL TRIAL: NCT07369882
Title: Comparison of Efficacy Between De-escalated Surgery and Standard Surgery After Neoadjuvant Immunotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma: A Randomized, Single-center Exploratory Clinical Study
Brief Title: Comparison of Efficacy Between De-escalated Surgery and Standard Surgery After Neoadjuvant Immunotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qunxing Li,MD (Other)
Responsible Party: Sponsor-Investigator, Qunxing Li,MD, MD PhD, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-990-01
Record Dates: First submitted 2025-12-31; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; locally advanced; De-escalated Surgery; Neoadjuvant
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Surgical De-escalation After Neoadjuvant Therapy
  Interventions: Procedure: Surgical De-escalation After Neoadjuvant Therapy
- Control arm (Active Comparator): Radical surgery combined with radiotherapy or chemoradiotherapy
  Interventions: Procedure: Radical surgery combined with radiotherapy or chemoradiotherapy

INTERVENTIONS:
Procedure: Radical surgery combined with radiotherapy or chemoradiotherapy — Radical resection of the primary tumor and neck dissection will be performed according to the NCCN guidelines, followed by adjuvant radiotherapy or chemoradiotherapy based on the postoperative pathological features.
  Arms: Control arm
Procedure: Surgical De-escalation After Neoadjuvant Therapy — The experimental group will undergo a de-escalated surgical approach, defined as follows:
  1. Primary tumor resection: The total diameter of the resection margins will be reduced by ≥30% compared with the pre-neoadjuvant therapy measurement. Resection will be performed with an additional 10-15 mm margin beyond the shrunken tumor boundary.
  2. Functional preservation: When appropriate, important anatomical structures and functional components such as the submandibular gland, mandible, epiglottis, oral commissure, parotid duct, eyeball, and major nerves may be preserved after thorough evaluation.
  3. De-escalated neck dissection:
  (1) Patients with clinically node-negative (cN0) neck status both before and after neoadjuvant immunotherapy will be exempted from neck dissection.
  (2) For midline-crossing lesions (e.g., tongue, hard palate, or soft palate), patients with contralateral clinically node-negative (cN0) neck status both before and after neoadjuvant immunotherapy will be exemp
  Arms: Experimental arm

SUMMARY:
This is a single-center, open-label, randomized, controlled, exploratory clinical trial designed to evaluate the efficacy and safety of de-escalated surgery compared with standard surgery in patients with resectable locally advanced head and neck squamous cell carcinoma (LA-HNSCC) who achieved a partial response (PR) or complete response (CR) after neoadjuvant immunochemotherapy. Eligible patients will be randomly assigned in a 1:1 ratio to either the de-escalated surgery group (experimental) or the standard surgery group (control). The de-escalated surgery group will undergo limited tumor resection and selective neck dissection based on clinical and imaging response, while preserving important anatomical structures and functions when feasible. The control group will receive standard surgical treatment following NCCN guidelines. All patients will be evaluated using RECIST 1.1 criteria for radiological response and will undergo enhanced CT or MRI at baseline, before the second cycle of neoadjuvant therapy, within one week before surgery, 30 days after surgery, and every 3 months thereafter until 2 years post-surgery, disease recurrence, death, or study completion. The study aims to assess whether de-escalated surgery can achieve similar oncologic outcomes while improving postoperative function and quality of life. The primary endpoints are disease-free survival (DFS), health-related quality of life (HRQoL), and 3- and 5-year overall survival rates (OS rate). A total of 60 patients will be enrolled over a 3-year period, with 30 in each group.

DETAILED DESCRIPTION:
This exploratory randomized controlled clinical study investigates the efficacy of de-escalated surgery versus standard surgery in patients with resectable locally advanced head and neck squamous cell carcinoma (LA-HNSCC) who have achieved partial response (PR) or complete response (CR) following neoadjuvant immunochemotherapy with a PD-1 inhibitor combined with nab-paclitaxel and carboplatin or cisplatin. The trial is designed to explore whether reducing the extent of surgical resection based on tumor response can maintain oncologic control while minimizing functional impairment.

Patients who meet the inclusion criteria will be randomized 1:1 into two groups. The experimental group will receive de-escalated surgery, including: (1) primary tumor resection with ≥30% reduction in the resection margin diameter compared to pre-neoadjuvant dimensions, with an additional 10-15 mm margin beyond the shrunken tumor boundary; (2) preservation of vital structures such as the submandibular gland, mandible, epiglottis, oral commissure, parotid duct, eyeball, and major nerves when appropriate; and (3) de-escalated neck dissection, exempting patients with cN0 status before and after therapy or limiting dissection in selected nodal levels. The control group will undergo standard surgery according to NCCN guidelines, including wide local excision of the primary tumor (10-15 mm margin) and comprehensive neck dissection.

Radiologic assessment will follow RECIST 1.1 using contrast-enhanced CT or MRI at multiple time points: baseline, prior to the second neoadjuvant cycle, within one week before surgery, 30 days postoperatively, and every three months up to 2 years or until recurrence, death, or study end. Baseline imaging will also rule out distant metastasis. Safety and postoperative follow-up will be conducted according to the same schedule.

The study's endpoints are disease-free survival (DFS), health-related quality of life (HRQoL), and overall survival rates (OS rate) at 3 and 5 years. The trial plans to recruit 60 patients over three years, with 30 assigned to each arm. Results from this study may provide clinical evidence for the feasibility of precision-based, response-adapted de-escalated surgery in head and neck squamous cell carcinoma management, potentially improving postoperative function and patient quality of life without compromising survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage III-IVa head and neck squamous cell carcinoma (HNSCC) according to the AJCC 8th edition TNM staging system, who have achieved a partial response (PR) or complete response (CR) after receiving neoadjuvant immunochemotherapy consisting of a PD-1 inhibitor in combination with nab-paclitaxel and carboplatin/cisplatin.
* No prior history of other malignant tumors.
* Aged between 18 and 75 years.
* Normal baseline (preoperative) clinical and laboratory findings:
* 1.Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L without the use of granulocyte colony-stimulating factor (G-CSF) within the previous 14 days
* 2.Platelet count ≥ 100 × 10⁹/L without blood transfusion within the previous 14 days
* 3.Hemoglobin > 9 g/dL without blood transfusion or erythropoietin use within the previous 14 days
* 4.Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
* 5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN
* 6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 mL/min
* 7. Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN
* 8. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. Subjects with TSH outside the normal range may be included if total T3 (or FT3) and FT4 are within normal limits
* 9. Normal myocardial enzyme profile (minor laboratory abnormalities judged by the investigator to be clinically insignificant are acceptable)
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to the first dose of study treatment (Cycle 1, Day 1). If the urine test is indeterminate, a serum test must be performed. Non-childbearing females are defined as those who have been postmenopausal for at least one year or have undergone surgical sterilization or hysterectomy.
* All subjects (male or female) with reproductive potential must agree to use highly effective contraception (annual failure rate <1%) during treatment and for at least 120 days after the last dose of study drug, or 180 days after the last dose of chemotherapy.
* Adverse events related to neoadjuvant therapy (e.g., bone marrow suppression, thyroiditis, hypothyroidism, hepatitis, nephritis, myocarditis, myositis, etc.) must have been adequately controlled and resolved to grade 0-2 before surgery. Patients assessed by anesthesiology as fit for general anesthesia may be included.
* Patients with pre-existing comorbidities prior to neoadjuvant therapy may also be enrolled if evaluated by anesthesiology and deemed able to tolerate general anesthesia.
* Signed written informed consent.

Exclusion Criteria:

* Diagnosis of another malignant tumor, or the primary lesion at the time of neoadjuvant therapy was not oral cancer.
* Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within 2 years prior to treatment. Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered systemic treatment.
* History of allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
* Known history of human immunodeficiency virus (HIV) infection (i.e., positive HIV-1/2 antibody).
* Untreated active hepatitis B infection, defined as HBsAg positivity with HBV-DNA levels exceeding the upper limit of normal (ULN) at the study site laboratory. Subjects meeting the following criteria may be enrolled:
* a. HBV viral load < 1000 copies/mL (200 IU/mL) prior to first dosing, provided antiviral therapy is administered throughout the study period to prevent viral reactivation
* b. Subjects who are anti-HBc(+), HBsAg(-), anti-HBs(-), and HBV-DNA(-) do not require prophylactic antiviral therapy but must undergo close monitoring for viral reactivation.
* Active hepatitis C virus (HCV) infection, defined as positive HCV antibody with detectable HCV-RNA above the lower limit of detection.
* Pregnant or lactating women.
* Presence of severe or uncontrolled systemic diseases, including but not limited to:
* 1. Cardiac disorders: severe arrhythmias (e.g., complete left bundle branch block, second-degree or higher atrioventricular block, ventricular arrhythmia, or persistent atrial fibrillation), unstable angina, or congestive heart failure (NYHA class ≥ II)
* 2. Vascular diseases: history of unstable angina, myocardial infarction, transient ischemic attack, or stroke within 6 months prior to enrollment
* 3. Poorly controlled hypertension: systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg
* 4. Pulmonary diseases: noninfectious pneumonitis requiring corticosteroid treatment within 1 year before first dosing, or active interstitial lung disease
* 5. Infectious diseases: active infections requiring systemic therapy, or severe uncontrolled infections
* 6. Active pulmonary tuberculosis
* 7. Gastrointestinal diseases: clinically active diverticulitis, intra-abdominal abscess, or intestinal obstruction
* 8. Hepatic disorders: liver cirrhosis, decompensated liver disease, or acute/chronic active hepatitis
* 9. Uncontrolled diabetes mellitus: fasting blood glucose (FBG) > 10 mmol/L
* 10. Renal dysfunction: urine protein ≥ ++ on routine urinalysis and 24-hour urinary protein > 1.0 g
* 11. Psychiatric disorders: severe mental illness that may affect treatment compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 2 years
  The time from randomization (or from the start of treatment in single-arm trials) to disease recurrence or death from any cause, whichever occurs first, will be analyzed. The Kaplan-Meier method will be used to estimate survival curves, and between-group comparisons will be performed using the log-rank test.
Change in Health-Related Quality of Life (HRQoL) Assessed by EORTC QLQ-C30 | Baseline (preoperative), 1 month after surgery, and at each follow-up visit (every 3 months up to 60 months).
  The EORTC QLQ-C30 is a validated, cancer-specific instrument developed by the European Organisation for Research and Treatment of Cancer (EORTC) to assess quality of life in cancer patients. It contains 30 items measuring global health status, functional domains (physical, role, cognitive, emotional, and social), and symptom scales (fatigue, pain, nausea/vomiting, etc.). Each item is scored on a 4-point Likert scale (1 = Not at all to 4 = Very much), except for two global health items scored from 1 (Very poor) to 7 (Excellent). Higher scores on functional and global health scales indicate better outcomes, whereas higher scores on symptom scales indicate worse outcomes.
Change in Head and Neck Cancer-Specific Quality of Life Assessed by EORTC QLQ-H&N43 | Baseline (preoperative), 1 month after surgery, and at each follow-up visit (every 3 months up to 60 months).
  The EORTC QLQ-H&N43 is a supplementary module to the QLQ-C30 designed to assess head and neck cancer-specific symptoms and functions. It includes 43 items covering domains such as pain, swallowing, speech, eating, social contact, and sexuality. Each item is rated on a 4-point Likert scale (1 = Not at all to 4 = Very much). Higher scores on symptom scales indicate worse symptoms or problems.

SECONDARY OUTCOMES:
Major pathological response | Perioperative
  MPR was assessed by two independent pathologists based on postoperative resection specimens, and discrepancies were resolved by a senior pathologist.
overall survival rate | 3 years and 5 years.
  Defined as the proportion of subjects who remain alive at 36 months from randomization or treatment initiation. For subjects lost to follow-up before death, the date of last contact will be considered as the censoring time.
Safety Endpoints | through study completion, an average of 1 year
  During the study and follow-up period, the severity of drug-related adverse events (DRAEs) and radiation-related adverse events was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, version 5.0). Surgery-related adverse events were classified based on the Clavien-Dindo grading system for surgical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Li, MD, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Raw data will not be publicly available. Aggregated and anonymized data may be shared upon reasonable request to the corresponding author after publication.